CLINICAL TRIAL: NCT01297049
Title: I-care: Stimulating Self-management in Patients With Type 2-diabetes Through Web-based Situational Feedback. A Pilot Study.
Brief Title: I-care: Stimulating Self-management in Patients With Type 2-diabetes
Acronym: I-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2010/427b
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Type 2; Obesity
Keywords: Diabetes; obesity; behavior therapy; self management
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Experimental)
  Interventions: Behavioral: Cognitive behavior therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavior therapy (CBT) — All patients will receive standard care (reassurance, education, physiotherapy, and necessary medication). Complementary to this standard care, the participants will be required to closely monitor their blood glucose levels, weight, eating behavior and daily activities, and to relay this information to the nurse specialist trained in treating somatic patients with CBT. The nurse will then suggest appropriate treatment decisions, the patients will receive situational feedback based on the electronic diary during 3 months (daily during 4 weeks intensive treatment and weekly during 2 months as a complement).
  Other Names: Life style counselling; Internet based counselling; Situational feedback

SUMMARY:
The overall objective of this pilot study is to develop a cost-effective treatment methodology delivered outside of traditional clinical setting, and based on modern technology for patients with diabetes type 2 also suffering from obesity. This study will investigate the feasibility of web based counselling and situational feedback through mobile supervising. The intention is to treat 10-15 patients. All participants will receive standard treatment delivered by their general practitioners. In addition the participants will fill in and send diaries to the supervisors each evening for 4 weeks reduced to a weekly frequency for the next two months period. The diary's schedule will be an evaluation of the day activities related to meals and food, medication management as well as the performed physical activities. The diary's schedule will also include blood glucose sample, and plans for the next day especially regarding physical activity. The participants will be able to view their own registrations on a web page. Daily/weekly situational feedback will be given to the participants within a cognitive behavioural framework to stimulate self-management. The primary outcome will be the HbA1c levels. Secondary outcomes will include evaluation of lifestyle outcomes such as physical activity levels and eating behaviour, and skills such as self-management of medication. In addition, the interventions effectiveness will examine mental health outcomes such as emotional distress and health-related quality of life.

DETAILED DESCRIPTION:
Diabetes and overweight have become a world health epidemic. The number of people suffering of these diseases is increasing due to population growth, aging, urbanization, and increasing prevalence of obesity and physical inactivity. The costs of diabetes affect health services, national productivity as well as individuals and families. Hospital in-patient costs for the treatment of complications are the largest single contributor to direct healthcare costs. Many of these complications and, therefore, their costs, are preventable. Intensive therapy, directed at the control of blood glucose, blood pressure etc, has been shown to be cost-effective in that, although initial costs are increased, it decreases longer term costs as a result of delayed or prevented complications . Diabetes self-management education is a multi-faceted process involving much more than helping people with diabetes to monitor their blood glucose, or take their medication as prescribed. Diabetes education must be an ongoing process rather than a one-time event because a person's health status and need for support change over time.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years old
* T2DM diagnosed > 3 months prior to study
* HbA1c 7,5-10%
* capability of filling in Norwegian questionnaires
* BMI ≥ 25
* able and willing to give signed informed consent
* willing to attend the full treatment schedule including ability to use mobile phones, computers and pocket computers

Exclusion Criteria:

* change in weight > 5kg during the last 3 months
* any mental or physical condition interfering with the protocol
* not having easy access to computers
* having reading problems

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-04; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose control with changes in Glycated hemoglobin (HbA1c) values | At the baseline and at the end of the intervention (3 months)
  HBA1c is a form of hemoglobin used primarily to identify the average plasma glucose concentration over prolonged periods of time. It is formed in a non-enzymatic glycation pathway by hemoglobin's exposure to plasma glucose. Normal levels of glucose produce a normal amount of glycated hemoglobin. As the average amount of plasma glucose increases, the fraction of glycated hemoglobin increases in a predictable way. This serves as a marker for average blood glucose levels over the previous months prior to the measurement

SECONDARY OUTCOMES:
Health Education Impact Questionnaire (heiQ); | At the baseline and after the end of the intervention (3 months)
  heiQ is a user-friendly instrument for the comprehensive evaluation of patient education programs with the following dimensions: positive and active engagement in life, health directed behavior, skill and technique acquisition, constructive attitudes and approaches, self-monitoring and insight, health service navigation, social integration and support, and emotional well-being.
Problem Areas in Diabetes (PAID) | At the baseline and after the end of the intervention (3 months)
  PAID is a brief self-report measure of diabetes-related distress that has been found to be useful in patients with diabetes (both type1 and 2). PAID scores have been found to show positive associations with HbA1c, and are a major predictor of poor adherence to treatment not involving general emotional distress
Food frequency questionnaire FFQ | At the baseline and after the end of the intervention (3 months)
  FFQ is a measure designed to measure average long-term diet or usual consumption with specified food items.
Audit of Diabetes Dependence Quality of Life (ADDQoL-19) | At the baseline and after the end of the intervention (3months)
  ADDQoL19 is a health-related quality of life questionnaire well designed to assess to what extent diabetes may affect different aspects of health related quality of life. The ADDQoL includes 2 introductory questions and 18 specific items, with the purpose of assessing, according to the patient's perspective, how much better his or her life would be if he/she did not have diabetes and how important each of these 19 aspects of life are for the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Andréa AG Nes, Mc, Principal Investigator — Oslo College University; Hilde Eide, Professor, Principal Investigator — Oslo College University/Buskerud College University
Locations (1):
- Oslo College University, Oslo, Arkeshus, Norway

REFERENCES:
- [Derived] Nes AAG, van Dulmen S, Brembo EA, Eide H. An mHealth Intervention for Persons with Diabetes Type 2 Based on Acceptance and Commitment Therapy Principles: Examining Treatment Fidelity. JMIR Mhealth Uhealth. 2018 Jul 3;6(7):e151. doi: 10.2196/mhealth.9942. PMID 29970357